CLINICAL TRIAL: NCT02950324
Title: Does Prehabilitation Improve Performance in Cardiopulmonary Exercise Testing and Reduce Insulin Resistance in Patients Undergoing Neo-adjuvant Treatment and Surgery for Oesophago-gastric Cancer?
Brief Title: Does Prehabilitation Improve Exercise Performance and Insulin Resistance After Surgery for Oesophago-gastric Cancer?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Sophie Allen, Research Fellow, Royal Surrey County Hospital NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16/LO/1702
Record Dates: First submitted 2016-10-13; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Cancer
Keywords: Prehabilitation; Oesophago-gastric; Cancer; Neo-adjuvant; Exercise; Cardiopulmonary exercise test; Insulin resistance
MeSH Terms: conditions — Neoplasms; Motor Activity; Insulin Resistance | interventions — Preoperative Exercise; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prehabilitation (Experimental): Patients in this (intervention) arm of the study will be enrolled into a multimodal programme that involves 15 weeks of exercise, nutritional support and psychological prehabilitation in the form of 'Medical Coaching'.
  Interventions: Behavioral: Prehabilitation
- Standard care (Active Comparator): Patients in the 'standard care' arm of the study will not receive the study intervention. The patients will continue to be offered the standard dietetic and psychological support as per the enhanced recovery pathway and current standard of care.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Prehabilitation — Patients in the intervention, 'Prehabilitation', arm of the study will be enrolled into a multimodal programme that involves 15 weeks of exercise, nutritional support and psychological prehabilitation in the form of 'Medical Coaching'. This will take place during neo-adjuvant treatment prior to oesophagectomy or gastrectomy for cancer.
  Arms: Prehabilitation
Behavioral: Standard care — Patients in the 'standard care' arm of the study will not receive the study intervention. The patients will continue to be offered theatients in this arm of the study will not receive the study intervention. The patients will continue to be offered the standard dietetic and psychological support as per the enhanced recovery pathway and current standard of care standard dietetic and psychological support as per the enhanced recovery pathway and current standard of care.
  Arms: Standard care

SUMMARY:
The purpose of this study is to evaluate the effect of a multimodal pre-operative prehabilitation programme during neo-adjuvant therapy on cardiopulmonary exercise performance and insulin resistance prior to resection for oesophago-gastric cancer.

DETAILED DESCRIPTION:
The trial objectives are as follows: Primary: To evaluate the effect of a prehabilitation programme during neo-adjuvant therapy on CPX performance prior to resection for oesophago-gastric cancer. Secondary: To investigate the impact of neo-adjuvant chemotherapy on insulin resistance; to determine whether a prehabilitation exercise programme is feasible during neo-adjuvant chemotherapy; to determine whether rehabilitation has a positive impact on quality of life outcomes; to investigate the impact of prehabilitation on clinical outcomes; to assess the effect of prehabilitation on nutritional status; to determine whether prehabilitation affects the stress response to surgery.

This study is a randomised controlled trial where patients will be stratified into 'fit' and 'unfit' groups based upon their anaerobic threshold and then randomised in a 1:1 ratio to receive multimodal prehabilitation or standard care prior to OG cancer surgery, during neo-adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients listed for elective oesophagectomy or total gastrectomy for cancer
* Must have capacity to consent
* Age 18-99

Exclusion Criteria:

* Known contraindication for CPX
* Physically unable to perform CPX test or undertake prehabilitation exercise programme
* Pregnant patients or those planning to become pregnant
* Lack of capacity to give informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change in cardiopulmonary exercise performance | Change in cardiopulmonary exercise performance between week 0 and week 17

SECONDARY OUTCOMES:
Change in insulin resistance | Change in insulin resistance between week 0 and week 17
Change in quality of life | Change in quality of life (as assessed by the EORTC QLQ C30 questionnaire) between week 0 and 6 months
Change in grip-strength | Change in grip-strength between 0 weeks and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Allen, MBBCh, Principal Investigator — Royal Surrey County Hospital NHS Trust
Locations (1):
- Royal Surrey County Hospital NHS Foundation Trust, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allen SK, Brown V, White D, King D, Hunt J, Wainwright J, Emery A, Hodge E, Kehinde A, Prabhu P, Rockall TA, Preston SR, Sultan J. Multimodal Prehabilitation During Neoadjuvant Therapy Prior to Esophagogastric Cancer Resection: Effect on Cardiopulmonary Exercise Test Performance, Muscle Mass and Quality of Life-A Pilot Randomized Clinical Trial. Ann Surg Oncol. 2022 Mar;29(3):1839-1850. doi: 10.1245/s10434-021-11002-0. Epub 2021 Nov 1. PMID 34725764
- [Derived] Allen S, Brown V, Prabhu P, Scott M, Rockall T, Preston S, Sultan J. A randomised controlled trial to assess whether prehabilitation improves fitness in patients undergoing neoadjuvant treatment prior to oesophagogastric cancer surgery: study protocol. BMJ Open. 2018 Dec 22;8(12):e023190. doi: 10.1136/bmjopen-2018-023190. PMID 30580268